CLINICAL TRIAL: NCT01997216
Title: Multifocal Lens Design Evaluation (US)
Brief Title: Multifocal Lens Design Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: C-12-036
Record Dates: First submitted 2013-11-19; First posted 2013-11-28 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2013-12

CONDITIONS: Refractive Error; Presbyopia
Keywords: contact lenses; multifocal
MeSH Terms: conditions — Refractive Errors; Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delefilcon A MF, then AOAMF (Other): Delefilcon A multifocal contact lenses, followed by lotrafilcon B multifocal contact lenses, as randomized. Each product was worn bilaterally (in both eyes) for 9 hours. The wear periods were separated by 2 ± 1 days.
  Interventions: Device: Delefilcon A multifocal contact lens; Device: Lotrafilcon B multifocal contact lens
- AOAMF, then Delefilcon A MF (Other): Lotrafilcon B multifocal contact lenses, followed by delefilcon A multifocal contact lenses, as randomized. Each product was worn bilaterally (in both eyes) for 9 hours. The wear periods were separated by 2 ± 1 days.
  Interventions: Device: Delefilcon A multifocal contact lens; Device: Lotrafilcon B multifocal contact lens

INTERVENTIONS:
Device: Delefilcon A multifocal contact lens — Investigational silicone hydrogel contact lens dispensed in low, medium, or high ADD per current AIR OPTIX® AQUA MULTIFOCAL fitting guidelines
Device: Lotrafilcon B multifocal contact lens — Commercially marketed silicone hydrogel contact lens dispensed in low, medium, or high ADD per current AIR OPTIX® AQUA MULTIFOCAL fitting guidelines
  Other Names: AIR OPTIX® AQUA MULTIFOCAL; AOAMF

SUMMARY:
The purpose of this study was to compare binocular high contrast, high illumination (HC/HI) visual acuity at near (40 centimeters) of new multifocal contact lenses against AIR OPTIX® AQUA MULTIFOCAL contact lenses when worn for 9 hours.

DETAILED DESCRIPTION:
Each participant was randomized to a specific sequence of lens wear, during which each lens type was worn bilaterally for 9 hours to compare performance characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Sign written Informed Consent document.
* Have spectacles that provide acceptable vision and be willing to wear them if unable to wear the study lenses.
* Be presbyopic with a spectacle add ≥ 0.50 diopter.
* Currently wearing soft contact lenses at least 5 days a week.
* Other protocol-specified inclusion criteria may apply

Exclusion Criteria:

* Eye injury or surgery within 12 weeks of enrollment in this trial.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in any clinical trial.
* Evidence of systemic or ocular abnormality, infection, or disease which is likely to affect successful wear of contact lenses (for at least 9 hours) or use of their accessory solutions as determined by the Investigator.
* Any use of medications for which contact lens wear could be contraindicated as determined by the Investigator.
* Binocular visual acuity worse than 20/25.
* Corrected by monovision.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Nick, Dipl.-Ing, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in the United States.
Pre-assignment Details: Of the 42 participants enrolled, 1 participant was exited as a screen failure and 1 participant was discontinued due to product unavailability prior to study product exposure. This reporting group includes all enrolled participants exposed to study product (40).
Period: First 9 Hours
Arm/Group | Delefilcon A MF, Then AOAMF | AOAMF, Then Delefilcon A MF
Started | 18 | 21
Completed | 18 | 21
Not Completed | 0 | 0
Period: Second 9 Hours
Arm/Group | Delefilcon A MF, Then AOAMF | AOAMF, Then Delefilcon A MF
Started | 19 (One participant was not exposed to Pair 1 due to product unavailability, but was exposed to Pair 2.) | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled participants exposed to study product.
Groups:
- Overall: Delefilcon A multifocal contact lenses and lotrafilcon B multifocal contact lenses, worn as randomized for 9 hours each.
Arm/Group | Overall
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Binocular HC/HI Visual Acuity at Near (40 cm)
Description: The participant read a Snellen chart at 40 centimeters with both eyes together while wearing study lenses. The Snellen acuity was converted into logMAR units (logarithm of the minimum angle of resolution). A 20/20 Snellen acuity equates to a logMAR acuity of 0.0 and is considered normal near eyesight. A negative logMAR value denotes better visual acuity.
Time Frame: Up to Hour 9
Population: All enrolled participants exposed to study product. 1 participant was not exposed to Delefilcon A MF due to product unavailability.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Delefilcon A MF: Delefilcon A multifocal contact lenses worn bilaterally (in both eyes) for 9 hours
- AOAMF: Lotrafilcon B multifocal contact lenses worn bilaterally (in both eyes) for 9 hours
Arm/Group | Delefilcon A MF | AOAMF
Number analyzed (Participants) | 39 | 40
logMAR
  Dispense (Hour 0) | 0.08 (0.10) | 0.06 (0.09)
  Hour 9 | 0.05 (0.08) | 0.05 (0.10)

2. Secondary Outcome: Mean Binocular HC/HI Visual Acuity at Distance
Description: The participant read a Snellen chart at a 20-foot equivalent distance with both eyes together while wearing study lenses. The Snellen acuity was converted into logMAR units (logarithm of the minimum angle of resolution). A 20/20 Snellen acuity equates to a logMAR acuity of 0.0 and is considered normal distance eyesight. A negative logMAR value denotes better visual acuity.
Time Frame: Up to Hour 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Delefilcon A MF | AOAMF
Number analyzed (Participants) | 39 | 40
logMAR
  Dispense (Hour 0) | -0.06 (0.04) | -0.06 (0.04)
  Hour 9 | -0.05 (0.08) | -0.05 (0.05)

3. Secondary Outcome: Mean Monocular Over-refraction (OR) at Distance
Description: OR is the amount of additional correction needed to improve visual acuity (VA). The OR at dispense was conducted with non-study product to determine lens power for the 9-hour wear. Dispensing of the study product (Pair 1 and Pair 2) was dependent upon lens power as determined by OR and resultant product availability. The OR at 9 hours was conducted with study product. All OR data is reported regardless whether study product was dispensed. Each eye contributed to the mean.
Time Frame: Up to Hour 9
Population: All enrolled participants exposed to study product. OR data is included for the 1 participant not exposed to Delefilcon A MF due to product unavailability.
Measure: Mean (Standard Deviation); unit: diopter
Arm/Group | Delefilcon A MF | AOAMF
Number analyzed (Participants) | 40 | 40
diopter
  Dispense (Hour 0) | 0.08 (0.14) | 0.06 (0.13)
  Hour 9 | 0.06 (0.13) | 0.03 (0.12)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (1 month). An Adverse Event (AE) was any untoward medical occurrence, unintended disease or injury, or untoward clinical sign whether or not related to the investigational medical device.
Description: This reporting group includes all enrolled participants exposed to study product. Exposure to the study product (Pair 1 and Pair 2) was dependent upon lens power as determined by OR and resultant product availability.
Arm/Group | Delefilcon A MF | AOAMF
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/39 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes